CLINICAL TRIAL: NCT04660630
Title: Real World Research Based on Genomics: Comparison of Precision and Experience Therapy for Chronic Cardiovascular and Cerebrovascular Diseases
Brief Title: A Real World Research: Comparison of Precision and Experience Therapy for Hypertension, Diabetes or Hyperlipidemias
Acronym: RCG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: China development research foundation (Unknown)
Responsible Party: Principal Investigator, Lihong Liu, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-1-21-1
Record Dates: First submitted 2020-11-19; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Hypertension,Essential; Diabetes type2; Hyperlipidemias
MeSH Terms: conditions — Essential Hypertension; Hyperlipidemias | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Precision group (Experimental): The subjects were tested for gene, and the corresponding therapeutic drugs were selected according to the results of gene detection. Regular follow-up was conducted according to the study design to evaluate the efficacy and adverse reactions.
  Interventions: Diagnostic Test: Gene detection of therapeutic drugs for chronic cardiovascular and cerebrovascular diseases; Behavioral: Regular follow-up and patient education
- Experience group (Active Comparator): The subjects were treated with drugs selected by doctors according to their experience. Follow up was performed at the same frequency as the precision group to evaluate the efficacy and adverse reactions.
  Interventions: Behavioral: Regular follow-up and patient education
- Observation group (No Intervention): The subjects did not accept any intervention, including follow-up, especially regular evaluation of efficacy and adverse reactions.

INTERVENTIONS:
Diagnostic Test: Gene detection of therapeutic drugs for chronic cardiovascular and cerebrovascular diseases — According to the results of drug gene chip detection, we combined with the clinical characteristics of the patient to choose more suitable cardiovascular and cerebrovascular treatment drugs.
  Other Names: Drug gene chip
  Arms: Precision group
Behavioral: Regular follow-up and patient education — The subjects received regular follow-up and patient education.
  Arms: Experience group; Precision group

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and health economics of precise drug use strategies based on pharmacogenomics compared with traditional drug use strategies for cardiovascular related chronic diseases.

DETAILED DESCRIPTION:
This study is a randomized controlled, single blind, multicenter clinical study. Beijing Chaoyang Hospital is the team leader, and director Liu Lihong is the project leader. The sub center is Daming County Street Town Health Center and Daming County Jiuzhi township health center. The team leader is responsible for the formulation, implementation and coordination of the research plan, and each sub center is responsible for the implementation of the specific study, patient management and research information feedback.

Three project groups were set up in this study: primary hypertension, type 2 diabetes and hyperlipidemia. In each group, the control group and the experimental group were set up, and the patients in two pilot towns of Daming County were selected by cluster stratified random sampling. The control group received the treatment of local researchers according to the traditional medication strategy. The patients in the experimental group were treated with the drug regimen formulated by local researchers according to the results of their pharmacogenomic test reports. The subjects were single blind.

ELIGIBILITY:
Inclusion Criteria:

1. They are 55 years old or above, with no gender restriction. They are permanent residents of Da-jie town and Jiu-zhi Township in Da-ming County.
2. Patients who meet one of the following:

   A. Hypertension project group:

   Primary hypertension was definitely diagnosed, systolic blood pressure ≥ 140 millimeter of mercury, diastolic blood pressure ≥ 90 millimeter of mercury, or both after drug treatment.

   B.Type 2 Diabetes project group:

   Patients with type 2 diabetes mellitus (non insulin dependent diabetes mellitus) who were diagnosed as type 2 diabetes mellitus (NIDDM) and had HbA1c ≥ 7.0% after drug treatment before enrollment.

   C.Hyperlipidemia project group:

   Those who were diagnosed as hyperlipidemia and were treated with or without medication before enrollment.
3. Patients who can provide real and reliable information related to drug treatment and efficacy evaluation

Exclusion Criteria:

1. Respondents who are not willing to fill in the true and reliable information form for any reason.
2. Patients with infectious diseases or serious life-threatening diseases such as malignant tumors.
3. Patients with severe liver and kidney function damage, affecting the choice of treatment drugs.
4. Patients with incomplete data related to study evaluation such as any of following:

A.The clinical data did not include systolic blood pressure, diastolic blood pressure, heart rate, glycosylated hemoglobin, fasting blood glucose, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglyceride core efficacy evaluation indicators.

B.The data related to adverse reactions required by clinical research can not be collected, including but not limited to the related drugs with adverse reactions, adverse reaction performance, time correlation, whether to stop suspicious drugs, and whether to stimulate adverse reactions by re-medication.

C.The information of medication compliance score and quality of life score could not be provided for any reason.

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
change of systolic pressure | 3 months
  Change of systolic blood pressure from baseline
change of diastolic pressure | 3 months
  Change of diastolic blood pressure from baseline
change of glycosylated hemoglobin | 3 months
  Change of glycosylated hemoglobin from baseline
change of fasting blood glucose | 3 months
  Change of fasting blood glucose from baseline
change of total cholesterol | 3 months
  Change of total cholesterol from baseline
change of low density lipoprotein cholesterol | 3 months
  Change of low density lipoprotein cholesterol from baseline
change of triglyceride | 3 months
  Change of triglyceride from baseline

SECONDARY OUTCOMES:
Compliance rate of blood pressure | 12 months
  Change of the compliance rate of blood pressure from baseline
Compliance rate of glycosylated hemoglobin | 12 months
  Change of the compliance rate of glycosylated hemoglobin from baseline
Compliance rate of low density lipoprotein cholesterol | 12 months
  Change of the compliance rate of low density lipoprotein cholesterol from baseline

OTHER OUTCOMES:
Change of the total costs of hypertension treatment | 12 months
  Change of annualized cost of hypertension treatment from baseline.
Change of the medicine costs of hypertension treatment | 12 months
  Change of annualized cost of hypertension treatment from baseline.
Change of the total costs of diabetes treatment | 12 months
  Change of annualized cost of diabetes treatment from baseline.
change of the medicine costs of diabetes treatment | 12 months
  Change of annualized cost of diabetes treatment from baseline.
Change of the total costs of hyperlipidemia treatment | 12 months
  Change of annualized cost of hyperlipidemia treatment from baseline.
Change of the medicine costs of hyperlipidemia treatment | 12 months
  Change of annualized cost of hyperlipidemia treatment from baseline.
Medication compliance | 12 months
  Change of the score of Morisky Medication Adherence Scale(MMAS-8) from baseline.
Health self assessment | 12 months
  Change of the score of EuroQol five dimensions questionnaire from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lihong Liu, Doctor, Principal Investigator — Beijing Chao Yang Hospital; Yue Qiu, Doctor, Principal Investigator — China development research foundation
Locations (1):
- Beijng Chao Yang Hospital, Beijing, China